CLINICAL TRIAL: NCT06657963
Title: Assessment of Opuntia Ficus-indica Supplementation on Improving Antioxidant and Inflammation Levels
Brief Title: Effects of Opuntia Ficus-indica Supplementation on Antioxidant Status and Inflammation Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeTree Asia Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LTA001
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Antioxidant Capabilities; Inflammation Biomarkers
Keywords: Antioxidant capabilities; Inflammation levels; Opuntia ficus-indica; Oral supplementation; Reactive Oxygen Species (ROS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental)
  Interventions: Dietary Supplement: Opuntia ficus-indica Supplementation

INTERVENTIONS:
Dietary Supplement: Opuntia ficus-indica Supplementation — Participants are required to consume oral supplementation of OFi fine powder packaged in individual sachets (LifeGreenTM, LifeTree Asia, Selangor, Malaysia) at the dosage of 1500 mg once daily for 3 months.

SUMMARY:
The goal of this clinical trial is to learn if supplementation Opuntia ficus-indica improve the antioxidant status and inflammation levels of the participants. The main questions it aims to answer are:

1. Does supplementation Opuntia ficus-indica improve the antioxidant status of the participants?
2. Does supplementation Opuntia ficus-indica improve the inflammation levels of the participants?

Researchers will compare before and after intervention to see if supplementation Opuntia ficus-indica works to improve the antioxidant status and inflammation levels of the participants.

Participants will:

Take drug supplementation Opuntia ficus-indica every day for 12 weeks. Visit the clinic once every 4 weeks for checkups and tests

DETAILED DESCRIPTION:
Study Design

This open-label, single-arm, prospective study involved a supplementation period of three months. The research was conducted in full compliance with the Declaration of Helsinki and the criteria outlined in Malaysian guidelines for Good Clinical Practice [76]. Participant eligibility was confirmed according to the protocol checklist, and written informed consent was obtained from all participants. The study received approval from the Institutional Ethics Committee, UCSI University, Malaysia, approval code is IEC-2022-FMHS-082.

Participants Selection

Participants were recruited through off-campus advertisements, and the study was conducted at UCSI University in Kuala Lumpur, Malaysia. The inclusion criteria were as follows: (1) generally healthy individually; (2) aged 18 years and above; (3) capable of understanding the study protocol and information; and (4) willing to provide informed consent. Exclusion criteria included: (1) currently undergoing supplementation aimed at enhancing antioxidant status, (2) having undergone major surgical procedures within six months before study entry and (3) pregnant or lactating woman. All participants were provided a participant information sheet and received a thorough explanation from the investigator. Written informed consent was obtained from each participant. Potential risks, including food allergies, were communicated to participants during the consent process.

Supplementation

Demographic characteristics and participants' medical histories were collected during the baseline visit. Afterwards, participants began daily oral supplementation of OFi fine powder packaged in individual sachets (LifeGreenTM, LifeTree Asia, Selangor, Malaysia) at the dosage of 1500 mg once daily for 3 months. The recommended intake dosage was communicated to participants upon their enrollment in the study. Participants prepared the beverages by mixing the contents of each sachet with 150 mL of lukewarm water and were instructed to consume it before meals. Three monthly follow-up visits were conducted. During each visit at weeks 0, 4, 8 and 12, a case report form (CRF) was utilized to gather information on vital signs, self-perceived general well-being and saliva samples for laboratory investigations. Participants were instructed to inform the research team immediately if they experienced adverse reactions to the tested supplement.

Laboratory Examinations Unstimulated saliva samples were collected using a sterile 2.0-mL vial. Participants uncapped the vial, placed the straw into the vial, and passively drooled down the straw for 90 secs. All samples were assayed for different parameters in duplicates. Total antioxidant capacity was assayed using Elabsciecne total T-AOC colourimetric assay kit (Elabscience Biotechnology Co. Ltd, Texas, United States), MDA as lipid peroxidation biomarker was assayed using Elabsciecne MDA colourimetric assay Kit (Elabscience Biotechnology Co. Ltd, Texas, United States), 3-NT as a biomarker of oxidative stress-derived protein damage was assayed using Elabsciecne 3-NT ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States) and 8-OHdG as a biomarker of oxidative stress-derived DNA damage was assayed using Elabsciecne 8-OHdG ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States). Inflammation levels were measured via IL-1beta, IL-6 and IL-10 biomarkers, using Elabsciecne ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States).

Vital Signs and General Wellbeing

Blood pressure and heart rate were measured using the Omron automatic blood pressure monitor HEM 7120 (Omron Healthcare, Kyoto, Japan). Temperature was measured using a Braun forehead infrared thermometer NTF 3000 (Braun GmbH, Kronberg, Germany). Visual Analogue Scale (VAS) was incorporated to self-evaluate their well-being. VAS is a psychometric instrument designed for participants to subjectively assess disease-related symptoms' severity or general well-being. It is a validated tool with demonstrated good validity and excellent reliability in evaluating general well-being and quality of life [35]. During the assessment, participants rated their condition on a 10-cm long horizontal VAS scale, where 0 points indicated the least healthy condition and 10 points indicated the most healthy condition.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy individually
* aged 18 years and above
* capable of understanding the study protocol and information
* willing to provide informed consent.

Exclusion Criteria:

* currently undergoing supplementation aimed at enhancing antioxidant status
* having undergone major surgical procedures within six months before study entry
* pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Antioxidant Status | From enrollment to the end of intervention at 12 weeks
  Unstimulated saliva samples were collected using a sterile 2.0-mL vial. Participants uncapped the vial, placed the straw into the vial, and passively drooled down the straw for 90 secs. All samples were assayed for different parameters in duplicates. Total antioxidant capacity was assayed using Elabsciecne total T-AOC colourimetric assay kit (Elabscience Biotechnology Co. Ltd, Texas, United States), MDA as lipid peroxidation biomarker was assayed using Elabsciecne MDA colourimetric assay Kit (Elabscience Biotechnology Co. Ltd, Texas, United States), 3-NT as a biomarker of oxidative stress-derived protein damage was assayed using Elabsciecne 3-NT ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States) and 8-OHdG as a biomarker of oxidative stress-derived DNA damage was assayed using Elabsciecne 8-OHdG ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States).
Inflammation Levels | From enrollment to the end of intervention at 12 weeks
  Unstimulated saliva samples were collected using a sterile 2.0-mL vial. Participants uncapped the vial, placed the straw into the vial, and passively drooled down the straw for 90 secs. All samples were assayed for different parameters in duplicates. Inflammatory markers IL-1beta, IL-6 and IL-10 were assayed using Elabsciecne ELISA Kit (Elabscience Biotechnology Co. Ltd, Texas, United States).

SECONDARY OUTCOMES:
Vital Signs - Blood Pressure | From enrollment to the end of intervention at 12 weeks
  Blood pressure were measured using the Omron automatic blood pressure monitor HEM 7120 (Omron Healthcare, Kyoto, Japan). The result is reported in the unit of millimeters of mercury (mmHg).
Vital Signs - Heart Rate | From enrollment to the end of intervention at 12 weeks
  Heart rate were measured using the Omron automatic blood pressure monitor HEM 7120 (Omron Healthcare, Kyoto, Japan). Heart rate is expressed as beats per minute (BPM).
Vital Signs - Body Temperature | From enrollment to the end of intervention at 12 weeks
  Temperature was measured using a Braun forehead infrared thermometer NTF 3000 (Braun GmbH, Kronberg, Germany). Body temperature is expressed in Celsius scale with the unit symbol °C.
General Wellbeing | From enrollment to the end of intervention at 12 weeks
  Visual Analogue Scale (VAS) was incorporated to self-evaluate their well-being. VAS is a psychometric instrument designed for participants to subjectively assess disease-related symptoms' severity or general well-being. It is a validated tool with demonstrated good validity and excellent reliability in evaluating general well-being and quality of life. During the assessment, participants rated their condition on a 10-cm long horizontal VAS scale, where 0 points indicated the least healthy condition and 10 points indicated the most healthy condition.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request. Additional documents including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following publication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available immediately following publication with no end date.
Access Criteria: Data will be shared with anyone who wishes to access with reasonable request.

REFERENCES:
- [Background] Martemucci G, Portincasa P, Di Ciaula A, Mariano M, Centonze V, D'Alessandro AG. Oxidative stress, aging, antioxidant supplementation and their impact on human health: An overview. Mech Ageing Dev. 2022 Sep;206:111707. doi: 10.1016/j.mad.2022.111707. Epub 2022 Jul 14. PMID 35839856